CLINICAL TRIAL: NCT06826794
Title: Frequency of Respiratory Acidosis in the Intensive Care Unit After Postoperative Cardiac Surgery. Impact of Using VentilO Application
Brief Title: VentilO Prospective Study
Acronym: VentilO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, François Lellouche, Principal investigator, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025-4300
Record Dates: First submitted 2025-01-28; First posted 2025-02-14 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Mechanical Ventilation Complication; Respiratory Acidosis
MeSH Terms: conditions — Acidosis, Respiratory | interventions — Nurse Clinicians

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinicians (Other): Clinicians include respiratory therapists, physcians, medical students
  Interventions: Other: Clinicians
- VentilO (Active Comparator): VentilO, smartphone application (or web plateform)
  Interventions: Device: VenitlO

INTERVENTIONS:
Other: Clinicians — Clinicians will determine respiratory parameters for mechanical ventilation upon arrival in the intensive care unit.
  Arms: Clinicians
Device: VenitlO — VentilO application (or web platerform) will determine respiratory parameters for mechanical ventilation upon arrival in the intensive care unit.
  Arms: VentilO

SUMMARY:
This is a randomized, open-label study comparing intial settings made by clinicians with settings recommandation made by the VentilO application immediately after intensive care unit admission.The study will allow direct comparison of the frequency of acidosis when patients are ventilated using the parameters of the VentilO application versus parameters chosen by the clinician. The variables determined by the clinician or VentilO will be respiratory rate, tidal volume and resulting minute ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years old)
* Intubated patients admitted to intensive care immediately post-operatively after cardiac surgery (all cardiac surgery combined)
* Ventilation in controlled mode (Assist Control or SIMV)

Exclusion Criteria:

* Absence of anthropometric data (height and weight) of patients available in the patient file
* Respiratory cycles mainly spontaneous on arrival
* Patient extubated on arrival in intensive care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Respiratory acidosis | 20 minutes after initiation of mechanical ventilation
  The frequency of respiratory acidosis on arterial gas after 20 minutes of mechanical ventilation (pH < 7.35 and PaCO2 > 45mmHg)

SECONDARY OUTCOMES:
Acid-base disorders on arrival in intensive care | 5 minutes after initiation of mechanical ventilation
  The frequency and severity of acid-base disorders on arrival in intensive care (pH<7.35 or pH > 7.45)

OTHER OUTCOMES:
Number of participants with hemodynamic shock - hypotension | Up to extubation
  Requiring >1L of volume repletion and/or use of amines at >0.05 mcg/kg/min or norepinephrine equivalent
Number of participants with a barotrauma | Up to extubation
  Presence of pneumothorax
Mortality | Up to intensive care unit discharge
  Intensive care unit mortality
Intensive care unit lenght of stay | Up to 28 days - intensive care unit length of stay - intensive care admission to intensive care discharge
  Intensive care unit lenght of stay
Number of participants with an acute kidney injury | Up to 28 days - intensive care unit length of stay - intensive care admission to intensive care discharge
  Acute kidney injury define by > 27 mmol for 48 hours or 1.5 x basline value (pre surgery)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No